CLINICAL TRIAL: NCT06191406
Title: Five-year Changes in Physical and Cognitive Function in Patients With Chronic Stroke: a Preliminary Retrospective Cohort Study
Brief Title: Five-year Changes in Patients With Chronic Stroke
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Yanisa Sinthunyathum, Resident in Physical medicine and rehabilitation department, Principal Investigator, Khon Kaen University
Other Study IDs: HE661406
Record Dates: First submitted 2023-12-09; First posted 2024-01-05 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Chronic Stroke
MeSH Terms: interventions — Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 6 minute walk test — Test for physical functions and cognitive functions
  Other Names: 10 meters walk test; Thai MMSE

SUMMARY:
Objective of the study:

* To determine changes in physical and cognitive function in patients with chronic stroke over 5 years
* To determine whether there are differences in physical and cognitive function in chronic stroke patients with different baseline levels of physical activity

ELIGIBILITY:
Inclusion Criteria:

- Stroke patients whose physical activity was assessed in 2018 - 2019 (Previous research study)

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stroke patients whose physical activity was assessed in 2018 - 2019 (Previous research study: Validity and Test-Retest Reliability of a Thai Stroke Physical Activity Questionnaire) which the population was stroke patients, aged ≥ 18 years with onset > 3 months. The study population is composed of patients who have achieved a compliance rate of more than 70% with the accelerometer within 1 week, total 50 people.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 5 years
  walk distance covered over a time of 6 minutes
10-meter walk test | 5 years
  comfortable & fast gait speed
Thai MMSE | 5 years
  test patient's cognition with mini-mental state examination (MMSE) Minimum score = 0 (worst outcome, poor cognitive function) Maximum score = 30 (better outcome, good cognitive function)

SECONDARY OUTCOMES:
Global quality of life | 5 years
  Global quality of life questionnaire which the patient will give their own score of their quality of life, scale from 0-100 (0 = worst quality of life, 100 = best quality of life)
Short FES-I | 5 years
  the Short Falls Efficacy Scale International (Short FES-I) questionnaire Minimum score = 7 (better outcome, less fear of falling) Maximum score = 28 (worst outcome, most fear of falling)
Fatigue assessment scale | 5 years
  Fatigue assessment scale questionnaire Minimum score = 10 (better outcome, less fatigue) Maximum score = 50 (worst outcome, more fatigue)
Barthel index | 5 years
  Barthel index questionnaire Minimum score = 0 (worst outcome, mostly dependent in daily living) Maximum score = 100 (better outcome, independent in daily living)

CONTACTS AND LOCATIONS:
Locations (1):
- Srinagarind Hospital Khon Kaen University, Khon Kaen, Thailand